CLINICAL TRIAL: NCT04961775
Title: Contrast Enhanced Ultrasound Using Sonazoid Diagnose Early Stage Endometrial Carcinoma
Brief Title: A Prospective Multi-center Study on Using Sonazoid Diagnose Early Stage Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Department of Interventional Ultrasound, Chinese PLA General Hospital
Other Study IDs: 2020-300-01-EC
Record Dates: First submitted 2020-11-16; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Endometrial Carcinoma Stage I
Keywords: Contrast Enhanced Ultrasound; Transvaginal ultrasound
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Injections; Sonazoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pathological diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Perflubutane Microspheres for Injection — 16 µL as perflubutane microbubbles (1 vial) is reconstituted with 2 mL of attached water for injection; usually, once for an adult, 0.015 mL/kg as dispersion is administered intravenously.
  Other Names: Sonazoid

SUMMARY:
Sonazoid as a new generation of ultrasound contrast agent.This study based on the features of Sonazoid specific angiography and higher mechanical index, the role of Sonazoid in the early diagnosis of Endometrial carcinoma was explored.

DETAILED DESCRIPTION:
Sonazoid is a second generation ultrasound contrast agent, which is composed of microbubbles containing chemically stable and insoluble Perfluorobutane (PFB) gas and a hard shell of phosphatidylserine sodium (2-3 μ m in diameter) wrapped in the outer layer. These microbubbles can generate stable nonlinear oscillations in a low-power acoustic field and generate echoes at the second harmonic frequency of the transmitted pulse for enhanced contrast harmonic imaging.

Because Sonazoid has the advantages of ultra long time development and good stability, Sonazoid has significant clinical advantages in the diagnosis of not focal liver lesions(FLLs) but breast tumor and other organ. However, there is no study based on contrast enhanced ultrasound(CEUS) using Sonazoid in early detection of Endometrial carcinoma. Therefore, based on the advantages of the new ultrasound contrast agent, using qualitative analysis and quantitative analysis method to collect large samples, compared with diagnosis results of standard reference, which has important clinical significance for early diagnosis, early detection and improving the accuracy of diagnosis of Endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients with Irregular Vaginal bleeding with endometrial thickness is greater than 5mm(Postmenopausal) or10mm (Premenopausal) via transvaginal ultrasound；
* 2)Able to perform curettage or other image examination and surgical pathological staging；
* 3) Patients with complete clinical data, pathological test and follow-up data；
* 4)Ability to understand, sign informed consent and agree to participate in the investigator.

Exclusion Criteria:

* 1)Patients without Endometrial carcinoma;
* 2)Women during pregnancy and lactation;
* 3)Those who are known to be allergic to ultrasound contrast agents;
* 4)Patients with arterial-venous (right to left) shunt in the heart or lung or with serious heart diseases or with serious lung diseases;
* 5)Any other condition makes patient not eligible for this clinical trial.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endometrial carcinoma who needs to biopsy or surgical resection;
Sampling Method: Probability Sample
Enrollment: 277 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of contrast-enhanced ultrasound in endometrial cancer by Sonazoid. | 10 months
  Pathology as a gold standard, to observe the diagnostic performance of Sonazoid in endometrial tumor:a prospective multicenter study based on quantitative and qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No